CLINICAL TRIAL: NCT00844532
Title: A Prospective, Non-randomized, 2 Arm (AP Arm & Omni-Link Elite [OE] Arm-separately Posted as: NCT01396525), Multi-center Clinical Trial to Evaluate the Safety and Efficacy of the Absolute Pro™ Peripheral Self-Expanding Stent System and the Omnilink Elite™ Peripheral Balloon-Expandable Stent System in Subjects With Atherosclerotic de Novo or Restenotic Lesions in the Native Common Iliac Artery and/or Native External Iliac Artery. CAUTION: The Omnilink Elite™ Peripheral Balloon-expandable Stent System is an Investigational Device. Limited by Federal (U.S.) Law to Investigational Use Only.
Brief Title: Trial to Evaluate the Safety & Efficacy of the Absolute Pro™ Peripheral Self-Expanding Stent System in Subjects With Atherosclerotic de Novo or Restenotic Lesions in the Native Common Iliac Artery and/or Native External Iliac Artery.
Acronym: MOBILITY AP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-107 Absolute Pro Arm (AP); 08-107 OE (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2009-02-12; First posted 2009-02-16 (Estimated); Results first posted 2012-09-07 (Estimated); Last update posted 2015-06-09 (Estimated); Status verified 2015-05

CONDITIONS: Peripheral Vascular Disease
Keywords: Atherosclerosis; Peripheral artery disease; Peripheral vascular disease; PAD; Claudication; Peripheral Arterial Occlusive Disease; Stent; PAOD; PVD
MeSH Terms: conditions — Peripheral Vascular Diseases; Atherosclerosis; Peripheral Arterial Disease; Intermittent Claudication; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Absolute Pro™ Peripheral Self-Expanding Stent System (Experimental): Arm includes both Absolute Pro™ and Absolute Pro™ Long Lesion (LL) Peripheral Self-Expanding Stent Systems
  Interventions: Device: Absolute Pro™ Peripheral Self-Expanding Stent System

INTERVENTIONS:
Device: Absolute Pro™ Peripheral Self-Expanding Stent System — Absolute Pro™ Peripheral Self-Expanding Stent System: Devices include both Absolute Pro™ and Absolute Pro™ LL Peripheral Self-Expanding Stent Systems. It is indicated for the treatment of a maximum of two bilateral de novo or restenotic atherosclerotic lesions in the native common iliac artery and/or native external iliac artery (one lesion per side).

SUMMARY:
To determine the safety and efficacy of the Absolute Pro™ Peripheral Self-Expanding Stent System in subjects with atherosclerotic de novo or restenotic lesions in the native common iliac artery and/or native external iliac artery.

ELIGIBILITY:
Clinical Inclusion Criteria:

1. Subject must be at least 18 and < 90 years of age.
2. Subject has been informed of the nature of the trial, agrees to its provisions, and has signed the informed consent form.
3. Subject must agree to undergo all protocol-required follow-up examinations and requirements at the investigational site.
4. History of symptomatic claudication (Rutherford Becker Clinical Category 2-3) or ischemic rest pain (Rutherford Becker Clinical Category 4).
5. Female subjects of childbearing potential must have had a negative pregnancy test before treatment, and must not be nursing at the time of treatment, and agree at time of consent to use birth control during participation in this trial up to and including the follow-up at 9 months.

Angiographic Inclusion Criteria

1. Up to two bilateral de novo or restenotic lesions of the native common iliac artery and/or native external iliac artery may be treated(one per side).
2. Common iliac artery lesion visually estimated to be ≥50% stenosis and ≤100% stenosis (total occlusion)
3. External iliac artery lesion visually estimated to be ≥50% stenosis and ≤99% stenosis
4. Lesion length for stenosis of the common or external iliac artery visually estimated to be ≥ 10 mm and ≤ 110 mm (Absolute Pro)
5. Lesion length for total occlusion of the common iliac artery visually estimated to be ≤40 mm
6. Target vessel reference diameter visually estimated to be ≥3.6 mm and ≤9.1 mm (Absolute Pro)
7. On the treatment side(s), patent superficial femoral and popliteal arteries and at least one patent distal outflow artery with in-line distal vessel flow to the foot as confirmed by arteriography. Patent is defined as < 50% stenosis.
8. Lesion length for stenosis of the common or external iliac artery visually estimated to be ≥ 10 mm and ≤ 50 mm (Omnilink Elite).
9. Target vessel reference diameter visually estimated to be ≥ 5.0 mm and ≤ 11.0 mm (Omnilink Elite).

Clinical Exclusion Criteria

1. Subject is unable to walk.
2. Subject has had recent major surgery (last 3 months) e.g., abdominal surgery, coronary artery bypass graft surgery, thoracic surgery.
3. Subject has received, or is on the waiting list for a major organ transplant (heart, lung, kidney, liver).
4. Subject is diagnosed as Rutherford Becker Clinical Category 0, 1, 5, or 6.
5. Subject has ulcers or lesions on the lower extremity(ies) of the target lesion side(s).
6. Subject has elevated serum creatinine > 2.0 mg/dl.
7. Subject has uncontrolled diabetes mellitus (DM) (serum glucose > 400 mg/dl).
8. Subject has had a myocardial infarction(MI)(Q-wave or NQWMI) within the previous 30 days.
9. Subject has had a stroke within the previous 30 days and/or has deficits from a prior stroke that limits the subjects ability to walk.
10. Subject has unstable angina defined as rest angina with ECG changes.
11. Subject has a groin infection, or an acute systemic infection that is currently under treatment.
12. Subject has acute thrombophlebitis or deep vein thrombosis in either extremity.
13. Subject requires any planned procedure within 30 days after the index procedure that would necessitate the discontinuation of aspirin, clopidogrel or ticlopidine following the procedure.
14. Subject has other medical illnesses (e.g., cancer or congestive heart failure) that may cause the subject to be non-compliant with protocol requirements, confound the data interpretation, or is associated with limited life-expectancy (i.e., less than 2 years).
15. Subject is currently participating in an investigational drug or device trial that has not completed the primary endpoint follow-up or that clinically interferes with the current trial endpoints.
16. Subject is unable to understand or unwilling to cooperate with trial procedures or is unwilling or unable to return to the treatment center for follow-up visits.
17. If intended stent is Absolute Pro, subject has known hypersensitivity or contraindication to nickel, titanium or platinum; subject has known hypersensitivity or contraindication to standard intraprocedure anticoagulant(s); subject has sensitivity to contrast which cannot be adequately pre-treated with medication.
18. Subject has known allergy or contraindication to aspirin or clopidogrel (Plavix®); if allergy or contraindication is to clopidogrel, subject is unable to tolerate ticlopidine (Ticlid®).
19. Subject has known bleeding disorder or hypercoagulable disorder, or will refuse blood transfusions.
20. Subject has suffered a gastrointestinal (GI) bleed within 30 days before the index procedure that would interfere with antiplatelet therapy.
21. If intended stent is Omnilink Elite, subject has known hypersensitivity or contraindication to cobalt chromium; subject has known hypersensitivity or contraindication to standard intraprocedure anticoagulant(s); subject has sensitivity to contrast which cannot be adequately pre-treated with medication.
22. Requirement of general anesthesia or spinal block for the procedure.
23. Presence of contralateral limb amputation that was performed to treat any non-traumatic disease in that limb, e.g. atherosclerotic, vascular, neuropathic.
24. Presence of bypass conduit in any outflow vessel, i.e. SFA, popliteal, anterior tibial, posterior tibial, peroneal, ipsilateral to the target lesion.
25. Subject requires a concomitant percutaneous endovascular procedure in another vessel, e.g. coronary.
26. Target lesion is in an iliac artery that has been previously stented.

Angiographic Exclusion Criteria

1. Subject has a totally occluded (100% stenosis) external iliac artery ipsilateral to the target lesion.
2. Subject has a totally occluded (100% stenosis) outflow artery (SFA) ipsilateral to the target lesion
3. Target lesion is within or adjacent to an aneurysm.
4. Lesion is located within or beyond a vessel that contains a bypass graft.
5. Lesion(s) requires atherectomy (or ablative devices) to facilitate stent delivery.
6. Subject has a history of aortic revascularization or has an abdominal aortic aneurysm > 3cm.
7. Lesion extends beyond the inguinal ligament.
8. Subject has angiographic evidence of thrombus in the target disease segment or vessel that is unresponsive to anti-thrombotic therapies.
9. Subject has multilevel disease in the target extremity that requires other staged procedures within 30 days before or after the procedure.
10. On the treatment side(s), subject is without patent superficial femoral and popliteal arteries and at least one patent distal outflow artery with in-line distal vessel flow to the foot as confirmed by arteriography. Patent is defined as < 50% stenosis.
11. Requirement for > 1 stent to treat full length of lesion.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-03; Primary Completion 2011-03 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony S. Das, MD, Principal Investigator — Presbyterian Heart Institute, Dallas, TX; Manish Mehta, MD, MPH, Principal Investigator — Albany Medical Center, Albany, NY.
Locations (1):
- Abbott Vascular, Santa Clara, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Trial population is comprised of male and female subjects with moderate to severe iliac artery atherosclerotic occlusive disease. Recruitment dates: March 23, 2009 through May 17, 2010
Groups:
- Absolute Pro™ Peripheral Self-Expanding Stent System: The Absolute Pro™ Peripheral Self-Expanding Stent System includes two versions of the device, the Absolute Pro™ and Absolute Pro™ Long Lesion (LL) Peripheral Self-Expanding Stent Systems, which are analyzed together per protocol pre-specification.
Period: Overall Study
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Started | 151
Completed | 112
Not Completed | 39
Not completed — Death | 16
Not completed — Withdrawal by Subject | 16
Not completed — Lost to Follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 85
  >=65 years | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 98
Region of Enrollment [Number; unit: participants]
  United States | 151

OUTCOME MEASURES:

1. Primary Outcome: Major Adverse Event (MAE) Rate
Description: Defined as death, myocardial infarction (MI), clinically-driven target lesion revascularization, and limb loss (major amputation only) on the treated side(s).
Time Frame: 9 months
Population: Intent to treat (ITT) population. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 147
percentage of participants | 6.1 [NA to 10.4] — One-sided 95% confidence interval was computed for this endpoint, lower bound is not provided.

2. Secondary Outcome: Device Success
Description: On a per device basis, the achievement of successful delivery and deployment of the trial device(s) at the intended location(s) and successful withdrawal of the delivery catheter(s).
Time Frame: acute: from beginning of index procedure to end of index procedure.
Population: Intent to treat (ITT) population. Included 192 study stents implanted plus 1 study stent inserted in subjects vasculature, but not implanted due to device malfunction. 1 study stent was excluded from device success because the chosen size was not appropriate, therefore the stent was not implanted.
Measure: Number (95% Confidence Interval); unit: percentage of devices
Units Other Than Participants: devices
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (devices) | 193
percentage of devices | 96.4 [92.7 to 98.5]

3. Secondary Outcome: Technical Success
Description: Technical success is defined, on per target lesion basis, device success and attainment of a final in-stent residual stenosis of < 30% by QA or as reported by the investigator, if QA is not available.
Time Frame: acute: from beginning of index procedure to end of index procedure.
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of target lesions
Units Other Than Participants: target lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (target lesions) | 181
percentage of target lesions | 87.3 [81.5 to 91.8]

4. Secondary Outcome: Procedure Success
Description: Procedure success is defined, per patient basis, as technical success without any of the following complications; death due to all causes, myocardial infarction (MI), major amputation of the treated limb(s), stent thrombosis and target lesion revascularization (TLR) within two (2) days after the index procedure or at hospital discharge, whichever is sooner.
Time Frame: Beginning of index procedure to 2 days post-index procedure or discharge, whichever is sooner
Population: ITT population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 85.4 [78.8 to 90.6]

5. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: The thigh brachial index is the ratio of the resting ipsilateral thigh systolic blood pressure as compared to the highest resting brachial systolic blood pressure. A normal range is 0.9 to 1.3.
Time Frame: Pre-procedure
Population: Per target limb analysis. ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 142
Number analyzed (Limbs) | 170
Ratio | 0.8 (0.2)

6. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: Post-procedure
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 136
Number analyzed (Limbs) | 162
Ratio | 1.0 (0.2)

7. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 1 month
Population: Per target limb analysis.ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 127
Number analyzed (Limbs) | 151
Ratio | 1.1 (0.2)

8. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 9 months
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 122
Number analyzed (Limbs) | 144
Ratio | 1.1 (0.2)

9. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 2 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 97
Number analyzed (Limbs) | 118
Ratio | 1.0 (0.2)

10. Secondary Outcome: Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 5
Time Frame: 3 years
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 92
Number analyzed (Limbs) | 109
Ratio | 1.1 (0.2)

11. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: The changes in thigh brachial index is the ratio of change between the pre-procedure measure and the stated timepoint measure.
Time Frame: Post-procedure
Population: ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 134
Number analyzed (Limbs) | 160
Ratio | 0.2 (0.2)

12. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 11
Time Frame: 1 month
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 122
Number analyzed (Limbs) | 145
Ratio | 0.3 (0.3)

13. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 11
Time Frame: 9 months
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 115
Number analyzed (Limbs) | 136
Ratio | 0.3 (0.2)

14. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 11
Time Frame: 2 years
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 92
Number analyzed (Limbs) | 112
Ratio | 0.2 (0.2)

15. Secondary Outcome: Changes in Thigh Brachial Index (TBI) for the Treated Limb(s)
Description: as for outcome 11
Time Frame: 3 years
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Ratio
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 86
Number analyzed (Limbs) | 102
Ratio | 0.2 (0.3)

16. Secondary Outcome: Walking Impairment Questionaire Scores
Description: Measured by the Walking Impairment Questionnaire (WIQ), a disease-specific instrument utilized to characterize walking ability through a questionnaire as an alternative to treadmill testing. It is a measure of subject-perceived walking performance for subjects with Peripheral Artery Disease (PAD) and/or intermittent claudication. The WIQ quantifies patient-reported walking speed, walking distance, and stair-climbing ability, respectively, on a scale of 0 (= worst) to 100 (= best).
Time Frame: Pre-procedure
Population: ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point.The highest possible score for each domain is 100%, which indicates no difficulty. Lowest possible score for each domain is 0%, which indicates inability to perform the activity.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
score on a scale
  Walking Distance Score | 14.0 (19.9)
  Walking Speed Score | 17.9 (20.8)
  Stair Climbing Score | 22.7 (23.9)

17. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 16
Time Frame: 1 month
Population: ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point.The highest score for each domain is 100%, which indicates no difficulty. Lowest possible score for each domain is 0%, which indicates inability to perform the activity.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 135
scores on a scale
  Walking Distance Score (N=134) | 53.8 (37.6)
  Walking Speed Score (N=135) | 51.8 (33.5)
  Stair Climbing Score (N=127) | 55.9 (36.7)

18. Secondary Outcome: Walking Impairment Questionaire Scores
Description: as for outcome 16
Time Frame: 9 months
Population: ITT population.The number of participants analyzed includes the subjects with available follow-up data at that time-point. The highest score for each domain is 100%, which indicates no difficulty.Lowest possible score for each domain is 0%, which indicates inability to perform the activity.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 127
scores on a scale
  Walking Distance Score (N=127) | 55.7 (39.6)
  Walking Speed Score (N=126) | 50.6 (33.9)
  Stair Climbing Score (N=119) | 59.2 (37.5)

19. Secondary Outcome: Walking Impairment Questionaire Scores
Description: Measured by the Walking Impairment Questionnaire (WIQ)
Time Frame: 2 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 99
scores on a scale
  Walking Distance Score (N=99) | 58.2 (37.1)
  Walking Speed Score (N=99) | 50.6 (32.4)
  Stair Climbing Score (N=95) | 59.1 (36.0)

20. Secondary Outcome: Walking Impairment Questionaire Scores
Description: Measured by the Walking Impairment Questionnaire (WIQ)
Time Frame: 3 years
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 94
scores on a scale
  Walking Distance Score (N=94) | 54.1 (40.0)
  Walking Speed Score (N=94) | 49.2 (33.0)
  Stair Climbing Score (N=88) | 58.9 (37.2)

21. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: The Rutherford Becker clinical category is a scale to measure chronic limb ischemia.
  Category and Clinical Description:
  0 = Asymptomatic, no hemodynamically significant occlusive disease, 1 = Mild claudication, 2 = Moderate claudication, 3 = Severe claudication, 4 = Ischemic rest pain, 5 = tissue loss, non-healing ulcer, or focal gangrene with diffuse pedal ischemia, 6 = Major tissue loss, extending above transmetatarsal level, functional foot no longer salvageable
Time Frame: Pre-Procedure
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
Percentage of Limbs
  0 | 0.0
  1 | 0.6
  2 | 28.2
  3 | 63.0
  4 | 8.3
  5 | 0.0
  6 | 0.0

22. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 1 month
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 134
Number analyzed (Limbs) | 161
Percentage of Limbs
  0 | 54.7
  1 | 26.7
  2 | 15.5
  3 | 2.5
  4 | 0.0
  5 | 0.6
  6 | 0.0

23. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 9 months
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 126
Number analyzed (Limbs) | 148
Percentage of Limbs
  0 | 60.1
  1 | 23.6
  2 | 14.2
  3 | 2.0
  4 | 0.0
  5 | 0.0
  6 | 0.0

24. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 2 years
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 98
Number analyzed (Limbs) | 119
Percentage of Limbs
  0 | 61.2
  1 | 25.6
  2 | 7.4
  3 | 4.1
  4 | 0.0
  5 | 1.7
  6 | 0.0

25. Secondary Outcome: Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 21
Time Frame: 3 years
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 95
Number analyzed (Limbs) | 113
Percentage of Limbs
  0 | 69.9
  1 | 18.6
  2 | 9.7
  3 | 1.8
  4 | 0.0
  5 | 0.0
  6 | 0.0

26. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: Change in Rutherford Becker Clinical Category:
  Worsening Rutherford Becker Clinical Category:
  Deterioration (an increase) in the Rutherford Becker Clinical Category by at least two categories from baseline and subsequently from the earliest post-procedural measurement or to a category 5 or 6.
  Improved Rutherford Becker Clinical Category:
  An improvement (a decrease) in the Rutherford Becker Clinical Category of at least one category from baseline and subsequently from the earliest post-procedural measurement.
Time Frame: Between baseline and 1 month
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 161
Percentage of Limbs
  Improved by >/= 3 categories | 42.2
  Improved by 2 categories | 30.4
  Improved by 1 category | 18.6
  No change | 8.1

27. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 26
Time Frame: Between baseline and 9 months
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 126
Number analyzed (Limbs) | 148
Percentage of Limbs
  Improved by >/= 3 categories | 47.3
  Improved by 2 categories | 29.1
  Improved by 1 category | 17.6
  No change | 6.1

28. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 26
Time Frame: Between baseline and 2 years
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 98
Number analyzed (Limbs) | 119
Percentage of Limbs
  Improved by >/= 3 categories | 52.9
  Improved by 2 categories | 19.8
  Improved by 1 category | 21.5
  No change | 3.3

29. Secondary Outcome: Changes From Baseline in Rutherford Becker Clinical Category for the Treated Limb(s)
Description: as for outcome 26
Time Frame: Between baseline and 3 years
Population: as for outcome 11
Measure: Number; unit: Percentage of Limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 95
Number analyzed (Limbs) | 113
Percentage of Limbs
  Improved by >/= 3 categories | 56.6
  Improved by 2 categories | 23.0
  Improved by 1 category | 15.0
  No change | 5.3

30. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: Target lesion revascularization was defined as any revascularization at the target lesion with or without evidence of target lesion diameter stenosis ≥ 50% determined by duplex ultrasonography (DUS) or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion).
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target lesions
  1 month | 100
  9 months | 95.6

31. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: Target lesion revascularization was defined as any revascularization at the target lesion with or without evidence of target lesion diameter stenosis ≥ 50% determined by DUS or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion).
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target lesions | 93.5

32. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: as for outcome 31
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesion
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesion) | 181
percentage of target lesions | 89.6

33. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Lesion Revascularization (TLR)
Description: as for outcome 31
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target lesions | 84.4

34. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years. Clinically-driven is defined as: Revascularization of the stent with evidence of new distal ischemic signs (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion, and target lesion diameter stenosis ≥ 50% determined by duplex ultrasound or arteriography.) (Note: This does not include coincidental overlap of a percutaneous transluminal angioplasty (PTA) balloon or stent into a study stent, that has <50% stenosis, while treating a non-target lesion in the target vessel).
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target lesions
  1 month | 100
  9 months | 97.1

35. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years. Clinically-driven is defined as: Revascularization of the stent with evidence of new distal ischemic signs (worsening Rutherford Becker Clinical Category that is clearly referable to the target lesion, and target lesion diameter stenosis ≥ 50% determined by duplex ultrasound or arteriography.) (Note: This does not include coincidental overlap of a PTA balloon or stent into a study stent, that has <50% stenosis, while treating a non-target lesion in the target vessel).
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target lesions | 94.7

36. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: as for outcome 35
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target lesions | 91.4

37. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Lesion Revascularization (CD-TLR)
Description: as for outcome 35
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects with target lesions who were event free at this timepoint.
Measure: Number; unit: percentage of target lesions
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target lesions | 86.9

38. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years. Target Vessel Revascularization (TVR) defined: Any revascularization of the target vessel, outside of the target lesion, with or without evidence of diameter stenosis ≥ 50% determined by DUS or arteriography, with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category that is clearly referable to the target vessel.)
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects with lesions in the target vessel who were event free at this timepoint.
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (lesions) | 181
percentage of target vessels
  1 month | 100
  9 months | 96.5

39. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 38
Time Frame: 18 months
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target vessels | 96.5

40. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 38
Time Frame: 2 years
Population: ITT population. This analysis represents those subjects with lesions in the target vessel who were event free at this timepoint.
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target vessels | 94.5

41. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Vessel Revascularization (TVR) for the Treated Limb(s)
Description: as for outcome 38
Time Frame: 3 years
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target vessels | 92.2

42. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Vessel Revascularization (CD-TVR) for the Treated Limb(s)
Description: Revascularization of the target vessel (outside the target lesion) with evidence of new distal ischemic signs (worsening Rutherford Becker clinical category that is clearly referable to the target vessel, and diameter stenosis ≥ 50% determined by DUS or arteriography).
Time Frame: 1 month and 9 months
Population: as for outcome 40
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target vessels
  1 month | 100
  9 months | 97.1

43. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Vessel Revascularization (CD-TVR) for the Treated Limb(s)
Description: as for outcome 42
Time Frame: 18 months
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target vessels | 97.1

44. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Vessel Revascularization (CD-TVR) for the Treated Limb(s)
Description: as for outcome 42
Time Frame: 2 years
Population: as for outcome 38
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target vessels | 95.1

45. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Clinically-driven Target Vessel Revascularization (CD-TVR) for the Treated Limb(s)
Description: as for outcome 42
Time Frame: 3 years
Population: as for outcome 40
Measure: Number; unit: percentage of target vessels
Units Other Than Participants: Lesions
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Lesions) | 181
percentage of target vessels | 94.3

46. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: Any revascularization of a target extremity vessel (distal to the superior border of the inguinal ligament on the ipsilateral side) with or without evidence of vessel diameter stenosis ≥ 50% determined by DUS or arteriography, and with or without new distal ischemic sign (worsening Rutherford Becker Clinical Category).
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects with vessels in the extremity with the target lesions, who were event free at this timepoint.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs
  1 month | 99.4
  9 months | 97.7

47. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: as for outcome 46
Time Frame: 18 months
Population: as for outcome 46
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs | 96.6

48. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: as for outcome 46
Time Frame: 2 years
Population: as for outcome 46
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs | 95.3

49. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Target Extremity Revascularization (TER) for the Treated Limb(s)
Description: as for outcome 46
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects with vessels in the extremity with the target lesions, who were event free at this timepoint.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs | 93.0

50. Secondary Outcome: Primary Stent Patency
Description: Absence of in-stent restenosis of the target lesion (≥50%) as determined by duplex ultrasound or angiogram and without interval reintervention since the initial study procedure.
Time Frame: 1 month
Population: ITT population. The number of participants analyzed includes the subjects with available follow-up data at that time-point.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 144
Number analyzed (Limbs) | 172
percentage of limbs | 98.3

51. Secondary Outcome: Primary Stent Patency
Description: as for outcome 50
Time Frame: 9 months
Population: as for outcome 50
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 130
Number analyzed (Limbs) | 154
percentage of limbs | 90.9

52. Secondary Outcome: Primary Stent Patency
Description: as for outcome 50
Time Frame: 2 years
Population: as for outcome 50
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 118
Number analyzed (Limbs) | 140
percentage of limbs | 80.7

53. Secondary Outcome: Primary Stent Patency
Description: as for outcome 50
Time Frame: 3 years
Population: as for outcome 50
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 106
Number analyzed (Limbs) | 125
percentage of limbs | 75.2

54. Secondary Outcome: Restenosis
Description: Defined as ≥ 50% stenosis at follow-up.
Time Frame: 9 months
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 130
Number analyzed (Limbs) | 154
percentage of limbs | 8.4 [4.6 to 14.0]

55. Secondary Outcome: Restenosis
Description: Defined as ≥ 50% stenosis at follow-up.
Time Frame: 2 years
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 116
Number analyzed (Limbs) | 136
percentage of limbs | 16.9 [11.0 to 24.3]

56. Secondary Outcome: Restenosis
Description: Defined as ≥ 50% stenosis at follow-up.
Time Frame: 3 years
Population: as for outcome 50
Measure: Number (95% Confidence Interval); unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 103
Number analyzed (Limbs) | 118
percentage of limbs | 20.3 [13.5 to 28.7]

57. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years
Time Frame: 1 month and 9 months
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants
  1 month | 100
  9 months | 96.1

58. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years
Time Frame: 18 months
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 94.5

59. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 92.3

60. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Death (All Cause)
Description: Outcome measure analysed at 1, 9 and 18 months, 2 and 3 years
Time Frame: 3 years
Population: ITT population. This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 88.3

61. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: The term myocardial infarction should be used when there is evidence of myocardial necrosis in a clinical setting consistent with myocardial ischemia.
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants
  1 month | 100
  9 months | 98.6

62. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: as for outcome 61
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 97.9

63. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: as for outcome 61
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 97.1

64. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Myocardial Infarction (MI)
Description: as for outcome 61
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 96.2

65. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: Amputation is defined as the removal of a body extremity by surgery. For this study, the definition of amputation will only include amputations of the limb(s) that was/were treated. A minor amputation will be defined as below the ankle; a major amputation will be defined as at or above the ankle.
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs
  1 month | 100
  9 months | 99.4

66. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: as for outcome 65
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs | 99.4

67. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: as for outcome 65
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs | 99.4

68. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Amputations (Major) of the Treated Limb(s)
Description: as for outcome 65
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects with target limbs who were event free at this time point.
Measure: Number; unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
Number analyzed (Limbs) | 181
percentage of limbs | 99.4

69. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: Embolism is the formation of a thrombus within the target lesion or stent with migration or atherosclerotic emboli migration to a distal artery.
Time Frame: 1 month and 9 months
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants
  1 month | 99.3
  9 months | 98.7

70. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: as for outcome 69
Time Frame: 18 months
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 98.7

71. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: as for outcome 69
Time Frame: 2 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 98.7

72. Secondary Outcome: Kaplan-Meier Estimate of Freedom From Embolic Events
Description: as for outcome 69
Time Frame: 3 years
Population: ITT population.This analysis represents those subjects who were event free at this time point.
Measure: Number; unit: percentage of participants
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 151
percentage of participants | 98.7

73. Secondary Outcome: Stent Thrombosis
Description: Stent thrombosis is defined as a total occlusion documented by DUS and/or arteriography at the stent site with or without symptoms that occurs ≤ 30 days post index procedure.
Time Frame: 1 month
Population: as for outcome 11
Measure: Number (95% Confidence Interval); unit: percentage of limbs
Units Other Than Participants: Limbs
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 148
Number analyzed (Limbs) | 177
percentage of limbs | 0.6 [0.0 to 3.1]

74. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: This measure indicates the absolute change between two timepoints represented by the mean.
  SF-12® Health Survey is validated measure using 12 questions to measure functional health and well-being from the patient's point of view. Scores on the scale are 0% (indicating poor perceived health status) to 100% (indicating excellent perceived health status) possible.
Time Frame: Baseline and 1 month
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 133
score on a scale | 9.9 (11.2)

75. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: as for outcome 74
Time Frame: Baseline and 9 months
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 124
scores on a scale | 9.5 (12.5)

76. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: as for outcome 74
Time Frame: Baseline and 2 years
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 101
scores on a scale | 10.0 (12.9)

77. Secondary Outcome: Changes in Quality of Life Measures: Physical Component Summary
Description: as for outcome 74
Time Frame: Baseline and 3 years
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 96
scores on a scale | 8.9 (11.6)

78. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 74
Time Frame: Baseline and 1 month
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 133
scores on a scale | 3.9 (10.9)

79. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 74
Time Frame: Baseline and 9 months
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 124
scores on a scale | 1.9 (10.4)

80. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 74
Time Frame: Baseline and 2 years
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 101
scores on a scale | 2.2 (13.4)

81. Secondary Outcome: Changes in Quality of Life Measures: Mental Component Summary
Description: as for outcome 74
Time Frame: Baseline and 3 years
Population: as for outcome 50
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Number analyzed (Participants) | 96
scores on a scale | 2.7 (12.4)

ADVERSE EVENTS:
Time Frame: 3 years
Description: Organ systems designations were chosen to match Abbott Categories coding as closely as possible and may differ from other coding systems. The number at risk excludes subjects who were lost to follow-up or withdrew from the study through 3 years without any events.
Arm/Group | Absolute Pro™ Peripheral Self-Expanding Stent System
Serious Adverse Events (participants affected / at risk) | 91/151
Other Adverse Events (participants affected / at risk) | 88/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Absolute Pro™ Peripheral Self-Expanding Stent System (N=151)
Bleeding (Injury, poisoning and procedural complications) | 1 (1) — Access Site Complication
Pain at insertion site (Injury, poisoning and procedural complications) | 1 (1) — Access Site Complication
Pseudoaneurysm (Injury, poisoning and procedural complications) | 1 (1) — Access Site Complication
Anemia (Blood and lymphatic system disorders) | 8 (9) — Blood Dyscrasia
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Blood Dyscrasia
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 9 (10)
Angina (Cardiac disorders) | 6 (6)
Arrhythmias (other than bradycardia) (Cardiac disorders) | 7 (7)
Bradycardia (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1)
Congestive Heart Failure (Cardiac disorders) | 6 (6)
Other: Chest Pain (Cardiac disorders) | 1 (1)
Other: Coronary Artery Disease (Cardiac disorders) | 7 (8)
Pain (Cardiac disorders) | 2 (2)
Surgery/Interventional Procedure (Cardiac disorders) | 2 (2)
Cardiac Arrest (Cardiac disorders) | 1 (1) — Cardiac/Hemodynamic
Hypertension (Cardiac disorders) | 1 (1) — Cardiac/Hemodynamic
Hypotension (Cardiac disorders) | 4 (4) — Cardiac/Hemodynamic
Syncope (Cardiac disorders) | 1 (1) — Cardiac/Hemodynamic
Abdominal Pain (Gastrointestinal disorders) | 1 (1)
Bleeding (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Gastrointestinal Bleed (Gastrointestinal disorders) | 6 (6)
Gastro-intestinal (Gastrointestinal disorders) | 2 (2)
Other: Cholecystitis (Gastrointestinal disorders) | 2 (2)
Other: Esophagitis (Gastrointestinal disorders) | 1 (1)
Other: Hernia (Gastrointestinal disorders) | 1 (1)
Other: Malnutrition (Gastrointestinal disorders) | 1 (1)
Other: Pancreatitis (Gastrointestinal disorders) | 1 (1)
Pain (Gastrointestinal disorders) | 1 (1)
Fever (Infections and infestations) | 1 (1)
Gastro-intestinal (Infections and infestations) | 1 (1)
Musculoskeletal (Infections and infestations) | 1 (1)
Other: Cellulitis (Infections and infestations) | 2 (2)
Other: Facial Abscess (Infections and infestations) | 1 (1)
Other: Foot Ulcer (Infections and infestations) | 1 (1)
Other: Inguinal Cellulitis (Infections and infestations) | 1 (1)
Other: Osteomyelitis (Infections and infestations) | 1 (1)
Other: Pancreatitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 9 (10)
Sepsis (Infections and infestations) | 3 (3)
Urinary Tract Infection (Infections and infestations) | 3 (4)
Viral, bacterial and fungal infections (Infections and infestations) | 1 (1)
Wound complication or wound infection (Infections and infestations) | 3 (4)
Diabetes (Metabolism and nutrition disorders) | 1 (1)
Other: Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Other: Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Genito-urinary (General disorders) | 2 (2) — Miscellaneous
Headache (General disorders) | 1 (1) — Miscellaneous
Musculoskeletal (General disorders) | 9 (11) — Miscellaneous
Other: Non Cardiac Chest Pain (General disorders) | 1 (1) — Miscellaneous
Surgery/Interventional Procedure (General disorders) | 2 (2) — Miscellaneous
Wound complication or wound infection (General disorders) | 1 (1) — Miscellaneous
Myocardial Infarction - Non-Q- wave (Cardiac disorders) | 1 (1)
Myocardial Infarction - Unknown (Cardiac disorders) | 3 (3)
Other: Non Stemi MI (Cardiac disorders) | 1 (1)
Confusion (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Mental Status Change (Nervous system disorders) | 2 (3) — Neurologic other than stroke
Myalgia (Nervous system disorders) | 1 (2) — Neurologic other than stroke
Other: Hydrocephalus (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Other: Anoxic Encephalopathy (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Other: Anxiety (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Other: Extremity Tremors (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Other: Metabolic Encephalopathy (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Other: Subarachnoid/Intracerebral Hemorrhage (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Seizure (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Surgery/Interventional Procedure (Nervous system disorders) | 1 (1) — Neurologic other than stroke
Transient Ischemic Attack (Nervous system disorders) | 2 (2) — Neurologic other than stroke
Dissection (Injury, poisoning and procedural complications) | 4 (4) — Procedure-related
Hypertension (Injury, poisoning and procedural complications) | 1 (1) — Procedure-related
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 4 (4) — Pulmonary
Other: Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Pulmonary
Renal Failure (Renal and urinary disorders) | 3 (4)
Other: Drug Toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory
Other: Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory
Other: Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Respiratory
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Respiratory
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 7 (7) — Respiratory
Other: cerebrovascular accident (Vascular disorders) | 2 (3) — Stroke
Other: Right Cerebellar Infarct (Vascular disorders) | 1 (1) — Stroke
Stroke: Unknown (Vascular disorders) | 2 (2)
Aneurysm (Vascular disorders) | 1 (1)
Dissection (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 2 (2)
Ischemia (Vascular disorders) | 1 (2)
Occlusion (Vascular disorders) | 9 (11)
Other: Carotid Stenosis (Vascular disorders) | 1 (1)
Other: Deep Vein Thrombosis (Vascular disorders) | 1 (1)
Other: Peripheral Vascular Disease (Vascular disorders) | 14 (25)
Pseudoaneurysm (Vascular disorders) | 1 (1)
Restenosis (Vascular disorders) | 6 (12)
Stenosis (Vascular disorders) | 21 (31)
Surgery/Interventional Procedure (Vascular disorders) | 2 (2)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Absolute Pro™ Peripheral Self-Expanding Stent System (N=151)
Arrhythmias (other than bradycardia) (Cardiac disorders) | 8 (8) — Cardiac
Hypotension (Cardiac disorders) | 10 (11) — Cardiac/Hemodynamic
Edema (non pulmonary) (General disorders) | 8 (9)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 53 (85)
Pain (General disorders) | 10 (11)
Other: Peripheral Vascular Disease (Vascular disorders) | 21 (26)
Stenosis (Vascular disorders) | 11 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days